CLINICAL TRIAL: NCT06731985
Title: The FAST- Study: The Follow-up After Shorter Tapes Study Effectiveness and Safety of Shorter Trans-obturator Tapes: A Prospective Observational Study From the Norwegian Female Incontinence Registry
Brief Title: The Follow-up After Shorter Tapes Study. Effectiveness and Safety of Shorter Trans-obturator Tapes.
Acronym: FAST
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Kjersti Rimstad, Doctor of Medicine, University Hospital, Akershus
Other Study IDs: FAST 2 and 3
Record Dates: First submitted 2024-12-02; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Stress Urinary Incontinence; Postsurgical Pain; Follow-Up Studies
Keywords: Long-term Follow-Up of shorter incontinence tapes
MeSH Terms: conditions — Urinary Incontinence, Stress; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women operated with shorter incontinence tapes: Women operated at AHUS between 2009 and 2020 for stress urinary incontinence with shorter incontinence tapes.

SUMMARY:
Urinary incontinence after pregnancy and labor affects 1 in 3 women and has a negative impact on quality of life (QOL), limiting women's physical activity and impairing sexual function. The traditional surgical method treating female urinary incontinence is to implant a sub-urethral synthetic sling, the currently preferred method in Norway. The majority of women treated with synthetic slings obtain great improvement in QOL, but a few experience severe complications including chronic pelvic pain. Several countries, therefore, have reverted to older, less effective surgical methods to avoid synthetic material. Awareness of severe complications has, in some Norwegian hospitals, led to a shift in technique towards shorter slings. With shorter slings, the goal is to achieve the same grade of continence as traditional slings, but with fewer serious complications. The long-term results and complications of these shorter slings are mostly unknown. Akershus University Hospital (AHUS) shifted to shorter slings early, in 2009, using a single incision mini-sling (SIMS) Ajust. Due to costs, AHUS changed to the intermediate sling TVT-O Abbrevo in 2016.

Through this study, we hope to establish if shorter slings have the same long-term results as traditional slings, and to investigate if shorter slings are safer than traditional slings, with less long-term complications, such as chronic pelvic pain. We plan to perform a long-term follow-up of women having had surgery with shorter slings at AHUS.

All patients operated with either SIMS Ajust or TVT-O Abbrevo at AHUS between 2009 and 2020 will be invited to a long-term follow-up. The study participants will be asked to fill in validated questionnaires regarding symptoms of urine leakage, QOL, any chronic pain related to the surgery, debut of pain, level of pain and any treatments for the pain. All women treated with the current used sling Abbrevo is invited to a physical examination including testing of their voiding function and a gynecologic examination to check for complications.

2D- and 3D ultrasound scans will be done on the TVT-O Abbrevo group to evaluate the position-, attachment- and any misplacement of the sling.

Women experiencing insufficient long-term results, such as chronic pain, will be offered a full examination and treatment.

DETAILED DESCRIPTION:
Background:

Stress Urinary incontinence (SUI) is a frequent consequence of childbirth and affects 1/3 of the general female population. It gravely diminishes the quality of life of numerous women by limiting their ability to be physically active, and impairing their sexual function. Mid-urethral sling (MUS) procedures have been the dominant surgical treatment for SUI over the last two decades. The traditional MUS procedures places a polypropylene mesh for support under the urethra, either in front of the bladder passing through the pelvis to the lower abdomen (tension free vaginal tape (TVT)), or to the side of the pelvis in the groin area (tension-free vaginal tape obturator inside-out (TVT-O)). These traditional techniques have well documented long lasting results and have improved the quality of life in most women with SUI. However, a few women experience serious complications such as severe chronic pain, dyspareunia, erosion/expulsion of the mesh, and voiding dysfunctions. Even though these devastating complications are rare, the consequence for affected women is lifelong reduced quality of life, even if the synthetic material is removed in its entirety. This has led to massive negative publicity, lawsuits against manufacturers and a movement in social media to ban these procedures. Several countries have therefore reverted to older, less effective surgical methods to avoid the use of synthetic materials.

Single incision mini-slings (SIMS), with much less synthetic mesh than traditional slings were introduced worldwide in 2006. In 2010, the TVT-O Abbrevo (TVT-A), an intermediate sling, was introduced hoping to refine the clinical performance of shorter slings. SIMS and intermediate slings have shown promising short-term results, but regarding long-term efficacy and complication rates, there are only a few published studies with small sample sizes. Given that shorter slings could represent a middle ground between the risk of severe complications and a loss of life quality due to untreated urinary incontinence, data on long-term effect and safety of the newer shorter slings is urgently needed. Retrieving such knowledge would make it possible to update surgical guidelines and provide patients considering surgical options with evidence-based recommendations.

Since 1998, Norway has had a compulsory registry of all incontinence surgeries performed in the country, the Norwegian Female Incontinence Registry (NFIR). Akershus University hospitals (AHUS) started already in 2009 using the SIMS Ajust and later intermediate slings as their preferred incontinence procedure. We therefore have a unique possibility to study the long-term results and complication rates by inviting women back to a long-term follow-up having undergone SIMS and intermediate sling surgery at AHUS. This follow-up also provides the possibility of investigating sling position using 2D dynamic and 3D trans-perineal ultrasound (TPUS). AHUS has the expertise in advanced ultrasound within the research group. How positioning of intermediate slings under the urethra may affect long-term success rates and adverse events is largely unknown. This lack of knowledge makes it difficult for gynecologists evaluating patients in need of repeat surgery, due to either treatment failure or long-term complications. Understanding the biomechanical effects visualized by ultrasound of the increasingly popular shorter slings would enable researchers and doctors to develop the treatment techniques for female incontinence further.

Research questions and methodology:

Part 2. Our over-all aim is to evaluate long-term subjective and objective outcomes of shorter slings.

Study design: Prospective observational study Long-term subjective outcomes Study population: Women treated with SIMS Ajust (n = 744) at Akershus University Hospital between 2009 and 2016 and Intermediate sling TVT-A (n= 318) at Akershus University Hospital between 2016 and 2020.

Follow-up: Potential study participants for both groups will be identified in the local quality database for female incontinence surgery (local NFIR) at AHUS and invited to a long-term follow-up (4-14 years) with questionnaires. The following questionnaires will be sent electronically to the patients together with study invitation and consent form: The validated NFIR questionnaire, the validated Pelvic Floor Impact Questionnaire (PFIQ-7) as well as additional questions regarding pain.

Primary outcomes: Long-term subjective cure rate. Secondary outcomes: Long-term treatment satisfaction scores, quality of life score and complication rates.

Long-term objective outcomes Study population: The 318 women having been treated with the currently most used shorter sling (TVT-A) at AHUS between 2016 and 2020 will be invited to a physical follow-up were they will undergo a clinical examination including assessment of objective cure, sling erosions and development of pelvic organ prolapse using the POP-Q system.

Primary outcomes: Long-term objective cure rates. Secondary outcomes: The same as defined under 1) Long-term subjective outcomes.

Part 3. We will study the positioning of the shorter sling TVT-A under the urethra using dynamic 2D and 3D ultrasound.

Our aim is to study the association between sling position, tension and anchoring under the urethra, and subjective and objective cure rate, and long-term complication rates, especially chronic pelvic pain.

Study design: Prospective observational study Study population: 318 women having had surgery with the intermediate sling TVT-A at AHUS between 2016 and 2020.

Follow-up: Women who consent to study participation and attend the physical follow-up will undergo a clinical examination that includes a transperineal ultrasound (TPUS) examination in the dorsal lithotomy position using a 3,5-6 MHz curved array abdominal probe. The TPUS volumes and images will be obtained with an empty bladder at rest and under full Valsalva.

Primary outcomes: Any association between sling position and subjective and objective cure rate and complication rates.

Secondary outcomes: Any association between sling position, tension or anchoring and long-term complications, especially chronic pelvic pain.

Statistics, power and sample size:

Part 2 This is a follow-up study of all women having been operated at AHUS with Ajust or TVT-A in the study period. Power calculations are not feasible as all women having had SIMS Ajust or TVT-A in the study period consenting to study participation will be analysed for subjective outcomes, whereas all women in the TVT-A group consenting to study participation will be analysed for objective outcomes.

Part 3 For the transperineal ultrasound (TPUS) we have estimated that a sample size of 107 is sufficient to draw valid conclusions. For further details on the calculation, please see the full Protocol.

Risk evaluation and countermeasures. The main risk to the project is patient inclusion. To get robust and valid scientific data we are depending on women being willing to participate in the project with clinical examinations and ultrasound measurements. We have estimated that a studyparticipation of 50% is sufficient to draw valid conclusion. For further information on this estimation please see the protocol

User Participation. The project has two user representatives. They have both participated in the planning of the project and given valuable comments in developing the study protocol. Both have agreed to stay on as part of the project group.

Ethical considerations: The Department Head at AHUS, the NFIR Management team, the NFIRs professional council, The Data Protection Officer at AHUS as well as the Regional Committee for Medical and Health Research Ethics in the Southeast of Norway (REC South East) has approved the study. Signed consent will be obtained from all study participants.

Study participants will only be examined using established techniques for the evaluation of women after incontinence surgery, the exception being the 3D ultrasound examination. None of them involves any additional risk for the participants.

Questionnaires and consent forms will be sent electronically and stored at the Services for Sensitive Data (TSD), as well as the research server at AHUS. Study participants who report persistent or recurring incontinence as well as any long-term complications related to the slings will be offered a full new clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* All women operated for stress-urinary incontinence with TVT-O Abbrevo of Ajust incontinence sling between 2009 and 2020.

Exclusion Criteria:

* Women operated with other incontinence operations or slings.

Ages: 25 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Female incontinence patients operated at AHUS between 2009 and 2021, aged between 25 and 90.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-05-18 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
NFIR questionnaire subjective cure rate | From 2009 to 2020 and evaluation in 2024
  Rate of subjective cure defined as a stress urinary incontinence index score <3 estimated by calculating a stress urinary incontinence index score from 4 clusters of questions in the NFIR questionnaire measuring degree of symptom bother from 0 to 12.
Objective cure rate on validated NFIR stress test | From 2009 to 2020 and evaluation in 2024.
  Objective cure defined as 0g leakage at a cough-jump pad weighing stress test.

SECONDARY OUTCOMES:
NFIR questionnaire quality of life score | From 2009 to 2020 and evaluation in 2024
  Level of quality of life score generated from 4 questions in the NFIR questionnaire measuring QoL impact. This index ranges from 0 (excellent quality of life) to 16 (poor quality of life).
Long-term complications | From 2009 to 2020 and evaluation in 2024.
  Rate of complications at long-term follow-up clinical examination.
NFIR treatment satisfaction rate | From 2009 to 2020 and evaluation in 2024.
  Rate of women answering "very satisfied with treatment" given the options "very satisfied", "moderately satisfied", "neither satisfied nor dissatisfied", "moderately dissatisfied" or "very dissatisfied" in the NFIR questionnaire.
NFIR total complication rate | From 2009 to 2020 and evaluation in 2024.
  Total complication rates in the NFIR questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Marie Ellstrom Engh Professor, PhD, Principal Investigator — Akershus university hospital HC
Locations (1):
- Akershus University Hospital, Lorenskog, Norway

IPD SHARING:
Plan to Share IPD: No
We will use anonymized data in our analysis.

REFERENCES:
- [Background] Ford AA, Rogerson L, Cody JD, Aluko P, Ogah JA. Mid-urethral sling operations for stress urinary incontinence in women. Cochrane Database Syst Rev. 2017 Jul 31;7(7):CD006375. doi: 10.1002/14651858.CD006375.pub4. PMID 28756647
- [Background] Ebbesen MH, Hunskaar S, Rortveit G, Hannestad YS. Prevalence, incidence and remission of urinary incontinence in women: longitudinal data from the Norwegian HUNT study (EPINCONT). BMC Urol. 2013 May 30;13:27. doi: 10.1186/1471-2490-13-27. PMID 23721491
- [Background] Ulmsten U, Henriksson L, Johnson P, Varhos G. An ambulatory surgical procedure under local anesthesia for treatment of female urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 1996;7(2):81-5; discussion 85-6. doi: 10.1007/BF01902378. PMID 8798092
- [Background] Delorme E, Droupy S, de Tayrac R, Delmas V. Transobturator tape (Uratape): a new minimally-invasive procedure to treat female urinary incontinence. Eur Urol. 2004 Feb;45(2):203-7. doi: 10.1016/j.eururo.2003.12.001. PMID 14734007
- [Background] Svenningsen R, Staff AC, Schiotz HA, Western K, Kulseng-Hanssen S. Long-term follow-up of the retropubic tension-free vaginal tape procedure. Int Urogynecol J. 2013 Aug;24(8):1271-8. doi: 10.1007/s00192-013-2058-2. Epub 2013 Feb 16. PMID 23417313
- [Background] Warro A, Ojala J, Ala-Nissila S, Laurikainen E. Nine years follow-up after TVT-O; the mesh still available for women suffering from urinary incontinence. J Gynecol Obstet Hum Reprod. 2023 Mar;52(3):102534. doi: 10.1016/j.jogoh.2023.102534. Epub 2023 Jan 13. PMID 36642377
- [Background] Schraffordt Koops SE, Bisseling TM, Heintz AP, Vervest HA. Quality of life before and after TVT, a prospective multicentre cohort study, results from the Netherlands TVT database. BJOG. 2006 Jan;113(1):26-9. doi: 10.1111/j.1471-0528.2005.00809.x. PMID 16398767
- [Background] Betschart C, Scheiner D, Hess E, Seifert B, Fink D, Perucchini D. Patient satisfaction after retropubic and transobturator slings: first assessment using the Incontinence Outcome Questionnaire (IOQ). Int Urogynecol J. 2011 Jul;22(7):805-12. doi: 10.1007/s00192-011-1366-7. Epub 2011 Feb 12. PMID 21318441
- [Background] Pace N, Artsen A, Baranski L, Palcsey S, Durst R, Meyn L, Moalli PA. Symptomatic improvement after mesh removal: a prospective longitudinal study of women with urogynaecological mesh complications. BJOG. 2021 Nov;128(12):2034-2043. doi: 10.1111/1471-0528.16778. Epub 2021 Jun 27. PMID 34047446
- [Background] Waltregny D, de Leval J. New surgical technique for treatment of stress urinary incontinence TVT-ABBREVO from development to clinical experience. Surg Technol Int. 2012 Dec;22:149-57. PMID 23109075
- [Background] Rudnicki M, von Bothmer-Ostling K, Holstad A, Magnusson C, Majida M, Merkel C, Prien J, Jakobsson U, Teleman P. Adjustable mini-sling compared with conventional mid-urethral slings in women with urinary incontinence. A randomized controlled trial. Acta Obstet Gynecol Scand. 2017 Nov;96(11):1347-1356. doi: 10.1111/aogs.13205. Epub 2017 Sep 15. PMID 28815547
- [Background] Alexandridis V, Rudnicki M, Jakobsson U, Teleman P. Adjustable mini-sling compared with conventional mid-urethral slings in women with urinary incontinence: a 3-year follow-up of a randomized controlled trial. Int Urogynecol J. 2019 Sep;30(9):1465-1473. doi: 10.1007/s00192-019-04004-w. Epub 2019 Jun 20. PMID 31222572
- [Background] Abdel-Fattah M, Cooper D, Davidson T, Kilonzo M, Boyers D, Bhal K, McDonald A, Wardle J, N'Dow J, MacLennan G, Norrie J. Single-incision mini-slings versus standard synthetic mid-urethral slings for surgical treatment of stress urinary incontinence in women: The SIMS RCT. Health Technol Assess. 2022 Dec;26(47):1-190. doi: 10.3310/BTSA6148. PMID 36520097
- [Background] Canel V, Thubert T, Wigniolle I, Fernandez H, Deffieux X. Postoperative groin pain and success rates following transobturator midurethral sling placement: TVT ABBREVO(R) system versus TVT obturator system. Int Urogynecol J. 2015 Oct;26(10):1509-16. doi: 10.1007/s00192-015-2723-8. Epub 2015 May 12. PMID 25963058
- [Background] Dyrkorn OA, Staff AC, Kulseng-Hanssen S, Dimoski T, Svenningsen R. The completeness and accuracy of the Norwegian Female Incontinence Registry. Acta Obstet Gynecol Scand. 2020 Dec;99(12):1618-1625. doi: 10.1111/aogs.13951. Epub 2020 Jul 20. PMID 32640493
- [Background] Shek KL, Dietz HP. Ultrasound imaging of slings and meshes in urogynecology. Ultrasound Obstet Gynecol. 2021 Apr;57(4):526-538. doi: 10.1002/uog.23545. PMID 33206433
- [Background] Dietz HP. Pelvic floor ultrasound: a review. Am J Obstet Gynecol. 2010 Apr;202(4):321-34. doi: 10.1016/j.ajog.2009.08.018. PMID 20350640
- [Background] Berild GH, Kulseng-Hanssen S. Reproducibility of a cough and jump stress test for the evaluation of urinary incontinence. Int Urogynecol J. 2012 Oct;23(10):1449-53. doi: 10.1007/s00192-012-1733-z. Epub 2012 Apr 19. PMID 22527539
- [Background] Hegde A, Nogueiras M, Aguilar VC, Davila GW. Dynamic assessment of sling function on transperineal ultrasound: does it correlate with outcomes 1 year following surgery? Int Urogynecol J. 2017 Jun;28(6):857-864. doi: 10.1007/s00192-016-3234-y. Epub 2016 Dec 26. PMID 28025681
- See also: FDA Public Health Notification: Serious Complications Associated with Transvaginal Placement of Surgical Mesh in Repair of Pelvic Organ Prolapse and Stress Urinary Incontinence — http://wayback.archive-it.org/7993/20170111190506/http://www.fda.gov/MedicalDevices/Safety/AlertsandNotices/PublicHealthNotifications/ucm061976.htm

DOCUMENTS (2):
  • Study Protocol (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT06731985/Prot_000.pdf
  • Informed Consent Form (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/85/NCT06731985/ICF_001.pdf